CLINICAL TRIAL: NCT03429621
Title: Effect of Simethicone on Reducing Bowel Interference During Minilaparotomy for Tubal Resection : a Randomized Controlled Trial
Brief Title: Effect of Simethicone on Reducing Bowel Interference During Tubal Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OBG-2560-05148
Record Dates: First submitted 2018-01-31; First posted 2018-02-12 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Sterility, Postpartum
MeSH Terms: conditions — Infertility, Female | interventions — Simethicone

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simethicone (Experimental): Each woman in the intervention group will be given Simethicone (Air-X®; 80 mg) 2 tablets chewing with water 50 ml at 2-8 hours before surgery.
  Interventions: Drug: Simethicone 80 MG
- No simethicone (No Intervention): The women will not be given Simethicone.

INTERVENTIONS:
Drug: Simethicone 80 MG — Simethicone (Air-X®; 80 mg) 2 tablets chewing with water 50 ml at 2-8 hours before surgery
  Arms: Simethicone

SUMMARY:
Tubal ligation is an everyday procedure for permanent female sterilization. It is usually performed after a vaginal delivery. Minilaparotomy is generally performed by doing small incision at infraumbilical area. This minimal access surgery requires adequate operative field exposure. Bowel interference, which obscures visualization of the operative field has been recognized as one of the major obstacles during this procedure. We found problems while doing surgery in small space and one of them is bowel interferance which obscures vision. This could lead to prolonged operation and complications. Simethicone is an antifoaming agent that use in bowel preparation prior to various procedures including laparoscopy, colonoscopy, endoscopy, and open major abdominal operations. Simethicone is proven to break the bubble and reduce intraluminal gas. This effect could result in reduction of bowel dilatation that interfere with the proper identification of the adnexal area. Benefit of taking simethicone prior to do minilaparotomy for tubal resection has not been examined.

Objectives: To examine the effect of simethicone on reducing bowel interference during minilaparotomy for tubal resection.

Design: A randomized controlled trial in women, age 20-45 years, undergoing postpartum sterilization after vaginal delivery at Faculty of Medicine, Chiang Mai University hospital. The participants will be randomly assigned into one of two study groups: intervention (taking simethicone) and control (not taking simethicone). For the intervention group, each woman will take simethicone (80 mg) 2 tablet chewing with water 50 ml at 2-8 hours before surgery. Fasting at least 6 hours before surgery. For the control group, the women will receive the same standard perioperative care without taking simethicone. The primary outcome measure will be surgeon-rated operative difficulty score, which is a visual analog scale based on assess from exposure of to the operative field in visual analog scale by surgeon. The secondary outcome will be operative time and incidence of intraoperative and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Women requesting postpartum sterilization by minilaparotomic tubal resection after vaginal delivery at Faculty of Medicine, Chiang Mai University

Exclusion Criteria:

* Pre-pregnancy BMI > 25 kg/m2
* Intraoperative general anesthesia or epidural anesthesia
* Previous abdominal surgery except for appendectomy
* Known bowel disorder including Crohn's disease, ulcerative colitis, previous bowel surgery

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Operative difficulty score | At the end of operation (within 1 hour after the completion of the operation)
  Operative difficulty scores will be assessed at the end of the operation by the operating surgeon. The surgeon will rate the difficulty of the operation from 0 to 10 according to the 10-cm visual analog scale with "0" represents the easiest operation and "10" represents the hardest operation.

SECONDARY OUTCOMES:
Operation time (Total) | From the start of skin incision creation to the completion of skin closure (up to 2 hours)
  The time duration from skin incision to completion of skin closure
Operation time (Intraabdominal) | From first entering abdominal cavity to start closing the abdominal peritoneum (up to 2 hours)
  The time duration from first entering abdominal cavity to start closing the abdominal peritoneum.

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Principal Investigator — Faculty of Medicine, Chiang Mai University
Locations (1):
- Department of OB-GYN, Faculty of Medicine, Chiang Mai University, Chiang Mai, Thailand